CLINICAL TRIAL: NCT06367413
Title: Effects of Whey Protein and N-acetylcysteine Co-ingestion on Skeletal Muscle Recovery Following Exercise-induced Muscle Damage.
Brief Title: Effects of Protein and NAC Co-ingestion on Skeletal Muscle Recovery
Acronym: PRoNAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Dimitrios Draganidis, Assistant Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTH-PRoNAC Study
Record Dates: First submitted 2024-04-07; First posted 2024-04-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Aseptic Muscle Injury
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, parallel group model.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, outcomes assessor and the principal investigator will be blinded until the intervention and the outcomes' assessment is done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants in this arm will execute 150 eccentric muscle contractions an receive a placebo supplement consisted of carbohydrate (maltodextrin).
  Interventions: Dietary Supplement: Placebo
- NAC (Experimental): Participants in this arm will execute 150 eccentric muscle contractions an receive a N-acetylcysteine supplement.
  Interventions: Dietary Supplement: NAC
- PRoNAC (Experimental): Participants in this arm will execute 150 eccentric muscle contractions an receive a supplement consisted of N-acetylcysteine and whey protein.
  Interventions: Dietary Supplement: NAC + Whey Protein

INTERVENTIONS:
Dietary Supplement: Placebo — Participants will receive three servings of carbohydrate per day during the 4-day experimental period. In specific, they will be supplemented with 0.31 gr of maltodextrin per kg of body weight in the first two servings (at mid-morning and mid-afternoon supplements) and with 0.49 gr of maltodextrin per kg of body weight in the pre-sleep serving (1.1 gr maltodextrin/kg BW/day).
  Arms: Placebo
Dietary Supplement: NAC — Participants will receive three servings of N-acetylcysteine per day during the 4-day experimental period. In specific, they will be supplemented with 13.33 mg of N-acetylcysteine per kg of body weight per serving (40 mg NAC/kg BW/day).
  Arms: NAC
Dietary Supplement: NAC + Whey Protein — Participants will receive three servings of N-acetylcysteine + whey protein per day during the 4-day experimental period. In specific, they will be supplemented with 0.31 gr of whey protein and 13.33 mg of N-acetylcysteine per kg of body weight in the first two servings (at mid-morning and mid-afternoon supplements) and with 0.49 gr of whey protein and 13.33 mg of N-acetylcysteine per kg of body weight in the pre-sleep serving (1.1 gr Whey protein + 40 mg NAC /kg BW/day).
  Arms: PRoNAC

SUMMARY:
Previous evidence suggests that though N-acetylcysteine (NAC) supplementation following eccentric exercise-induced muscle damage disrupts the skeletal muscle's repair and remodelling process at 8 days of recovery, it attenuates substantially the decline of skeletal muscle performance during the first 48 hours of recovery. The enhanced performance capacity during the first phase of recovery in response to NAC supplementation might be attributed to the altered redox status in skeletal muscle as a consequence of the NAC-mediated elevation of reduced glutathione (GSH) levels. The rise in GSH results in a redox-dependent attenuation of immune cell mobilisation and reduction of oxidative stress response, leading to a blunted rise of muscle damage and inflammatory markers during the first 2-3 days of recovery. However, following exercise-induced muscle damage, protein synthesis increases in skeletal muscle over the next 24-48 hours to support its repair process, and thus protein supplementation might accelerate the recovery process by enhancing the protein synthetic response. Therefore, the present study aims at investigating for first time the combined effect of NAC and whey protein supplementation on the short-term (during the first 72 hours) recovery process of skeletal muscle following damaging exercise (eccentric exercise) and compared it with the well-documented efficacy of NAC supplementation. The results of this study might be particularly useful for athletes, such as those in soccer and basketball, that participate in 3 games or intense training sessions during the same macrocycle with only 48-72 hours of recovery in-between.

DETAILED DESCRIPTION:
Participants will initially undergo baseline testing including assessment of their (i) anthropometrics, (ii) body composition via DXA, (iii) habitual physical activity level via accelerometry, (iv) resting metabolic rate via indirect calorimetry, (v) daily dietary intake via 7-day dietary recalls and (vi) cardiorespiratory fitness using a treadmill ramp test. After baseline testing, participants will be assigned to (a) a Placebo, (b) a N-acetylcysteine (NAC) or (c) a N-acetylcysteine + Whey protein (PRoNAC) group, in a randomized, double-blind, placebo-controlled, parallel group, repeated measures design. In all groups, participants will execute an eccentric exercise protocol on an isokinetic dynamometer consisted of 150 eccentric muscle contractions. Before exercise as well as at 1-, 2-, 3-, 24-, 48- and 72-hours post-exercise they will undergo assessment of their maximal voluntary isometric peal torque, maximal countermovement jump height and muscle soreness level. In addition, blood sample will be drawn before exercise and at 24-, 48- and 72-hours post-exercise for the determination of myoglobin concentration, reduced (GSH) and oxidized (GSSG) glutathione content, protein carbonyl formation and catalase activity.

Throughout the 4-day experimental period (Day 1: exercise day, Days 2, 3 and 4: 24-, 48- and 72-hours post-exercise, respectively) participants will receive daily, 3 doses from the respective supplement as follows: the 1st dose at mid-morning (between breakfast and lunch), the 2nd dose at mid-afternoon (post-exercise on day 1 and between lunch and dinner on days 2-4) and the 3rd dose before sleep. In Placebo group, participants will be supplemented with 0.31 gr of maltodextrin per kg of body weight in the first two servings (at mid-morning and mid-afternoon supplements) and with 0.49 gr of maltodextrin per kg of body weight in the pre-sleep serving (1.1 gr maltodextrin/kg BW/day). In NAC group, participants will be supplemented with 13.33 mg of N-acetylcysteine per kg of body weight per serving (40 mg NAC/kg BW/day). In PRoNAC group participants will be supplemented with 0.31 gr of whey protein and 13.33 mg of N-acetylcysteine per kg of body weight in the first two servings (at mid-morning and mid-afternoon supplements) and with 0.49 gr of whey protein and 13.33 mg of N-acetylcysteine per kg of body weight in the pre-sleep serving (1.1 gr Whey protein + 40 mg NAC /kg BW/day).

ELIGIBILITY:
Inclusion Criteria:

* Free of asthma, kidney disease, bleeding disorders, peptic ulcers.
* Free of musculoskeletal injuries and limitations.
* Abstain from dietary energy restriction.
* Do not use medication such as anti-inflammatory drugs, antibiotics, antihypertensive drugs or anticoagulants.
* Do not use dietary supplements such as protein, carbohydrate, antioxidants, vitamins etc.
* Free of N-acetylcysteine intolerance.
* Non-smokers.
* Abstain from alcohol throughout the study.

Exclusion Criteria:

* Presence of asthma, kidney disease, bleeding disorders, peptic ulcers.
* Musculoskeletal injuries and limitations.
* Dietary energy restriction.
* Use of anti-inflammatory drugs, antibiotics, antihypertensive drugs or anticoagulants.
* Use of dietary supplements such as protein, carbohydrate, antioxidants, vitamins etc.
* N-acetylcysteine intolerance.
* Smoking.
* Alcohol consumption during the study.

Ages: 18 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in maximal voluntary isometric muscle contraction. | Before exercise and at 1-, 2-, 3-, 24-, 48- and 72-hours post-exercise.
  Maximal voluntary isometric muscle contraction will be assessed on an isokinetic dynamometer.
Change in countermovement jump height. | Before exercise and at 1-, 2-, 3-, 24-, 48- and 72-hours post-exercise.
  Countermovement jump height will be assessed by using the Optojump Next system.
Change in delayed onset of muscle soreness (DOMS) | Before exercise and at 1-, 2-, 3-, 24-, 48- and 72-hours post-exercise.
  DOMS of the knee extensors of the dominant limb will be evaluated by palpation of the relaxed muscle's belly and distal region with participants rating the perceived soreness on a visual analogue scale ranging from 1 to 10.
Change in reduced glutathione content. | Before exercise and at 24-, 48- and 72-hours post-exercise.
  Reduced glutathione content in blood erythrocytes will be assessed using spectrophometric method.
Change in oxidized glutathione content. | Before exercise and at 24-, 48- and 72-hours post-exercise.
  Oxidized glutathione content in blood erythrocytes will be assessed using spectrophometric method.
Change in catalase activity. | Before exercise and at 24-, 48- and 72-hours post-exercise.
  Catalase activity will be measured spectrophotometrically in red blood cells.
Change in protein carbonyl concentration | Before exercise and at 24-, 48- and 72-hours post-exercise.
  Protein carbonyl concentration will be measured spectrophotometrically in red blood cells.
Change in myoglobin concentration in blood. | Before exercise and at 24-, 48- and 72-hours post-exercise.
  Myoglobin concentration in blood will be assessed using an automatic biochemistry analyzer and commercially available kits.

SECONDARY OUTCOMES:
Participants' lean body mass | At baseline.
  Lean body mass (kg) will be assessed using dual-energy X-ray absorptiometry (DXA) instrumentation.
Participants' daily physical activity-related energy expenditure. | At baseline.
  Physical activity-related energy expenditure (kcal/day) will be assessed using accelerometers.
Participants daily dietary intake. | At baseline.
  Daily dietary intake composition (total kcal/day, gr of protein, gr of CHO and gr of fat intake/day, gr/mg of micronutrient intake/day) will be monitored using 24-h dietary recalls that will be analyzed by a trained dietitian using a dietary analysis software.
Participants' resting metabolic rate. | At baseline.
  Resting metabolic rate will be assessed using indirect calorimetry.
Participants' cardiorespiratory fitness status. | At baseline.
  Cardiorespiratory fitness will be assessed using a treadmill ramp test.
Participants' fat free mass. | At baseline.
  Fat free mass will be assessed using dual-energy X-ray absorptiometry (DXA) instrumentation.
Participants' fat mass. | At baseline.
  Fat mass will be assessed using dual-energy X-ray absorptiometry (DXA) instrumentation.
Participants' body fat percent. | At baseline.
  Body fat percent (%) will be assessed using dual-energy X-ray absorptiometry (DXA) instrumentation.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Draganidis, PhD, Principal Investigator — University of Thessaly, Department of Physical Education and Sport Science
Locations (1):
- Department of Physical Education and Sport Science, University of Thessaly, Trikala, Karies, Greece